CLINICAL TRIAL: NCT06838975
Title: Effectiveness of Virtual Reality Rehabilitation to Improve Cognitive, Emotional, Relational, and Motor Domains in Patients With Neurological and Neurodegenerative Disorders
Brief Title: Virtual Reality Rehabilitation for Cognitive, Emotional, and Motor Recovery in Neurological Disorders
Acronym: NeuroVR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Maria Grazia Maggio, PhD, PsyD, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEURO_VR; Current Research Funds 2025 (Other Grant/Funding Number: Ministry of Health Italy)
Record Dates: First submitted 2025-01-31; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Acquired Brain Injuries; Spinal Cord Injury; Multiple Sclerosis; Parkinson Disease
Keywords: Neurorehabilitation; Virtual Reality; Cognitive and motor recovery; cognitive rehabilitation; neurological disorders
MeSH Terms: conditions — Spinal Cord Injuries; Multiple Sclerosis; Parkinson Disease; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: This study follows a randomized controlled trial (RCT) design with a parallel assignment model, where participants are randomly allocated to either a VR-based rehabilitation group or a traditional rehabilitation control group. The intervention consists of 20 sessions over 8 weeks, with follow-up assessments at post-intervention (T1) and 3 months (T2). Blinded evaluators will conduct neurological, cognitive, motor, and neurophysiological assessments (EEG, MRI, fNIRS, motion analysis) at each time point. This model allows for a rigorous comparison of VR rehabilitation with conventional therapy, examining its effects on functional recovery, neurophysiological changes, and treatment adherence.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: This study uses a single-blind design, where outcome assessors are masked to group assignments to reduce bias. Participants and therapists delivering the intervention are aware of the assignment due to the nature of the rehabilitation protocols, but the neuropsychological, motor, and neurophysiological evaluations (EEG, MRI, motion analysis) will be conducted by blinded assessors who do not know whether the participant belongs to the VR Training Group or the Active Control Group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Training Group (Experimental): Participants in the VR Training Group will undergo a virtual reality-based rehabilitation program designed to improve cognitive, emotional, social, and motor functions. The intervention consists of 20 sessions over 8 weeks (3 sessions per week), using immersive and non-immersive VR systems tailored to individual needs. The program integrates interactive exercises, real-time feedback, and task-oriented training to enhance motor function, cognitive abilities, and patient engagement. Neurophysiological changes will be monitored through EEG, MRI, and motion analysis to assess brain plasticity and functional improvements.
  Interventions: Device: VR Training
- Active Control Group (Active Comparator): Participants in the Active Control Group will receive traditional cognitive and motor rehabilitation following standard clinical practices. The intervention consists of 20 sessions over 8 weeks (3 sessions per week), focusing on conventional physical therapy, cognitive training, and task-oriented exercises to enhance motor function and cognitive abilities. This group serves as a comparison to evaluate the effectiveness of VR-based rehabilitation. Neurophysiological changes will be monitored using EEG, MRI, and motion analysis to assess functional improvements.
  Interventions: Other: traditional cognitive and motor rehabilitation following standard clinical practices

INTERVENTIONS:
Device: VR Training — Participants in the VR Training Group will undergo a virtual reality-based rehabilitation program designed to improve cognitive, emotional, social, and motor functions. The intervention consists of 20 sessions over 8 weeks (3 sessions per week), using immersive and non-immersive VR systems tailored to individual needs. The program integrates interactive exercises, real-time feedback, and task-oriented training to enhance motor function, cognitive abilities, and patient engagement. Neurophysiological changes will be monitored through EEG, MRI, and motion analysis to assess brain plasticity and functional improvements.
  Other Names: Experimental Group
  Arms: VR Training Group
Other: traditional cognitive and motor rehabilitation following standard clinical practices — Participants in the Active Control Group will receive traditional cognitive and motor rehabilitation following standard clinical practices. The intervention consists of 20 sessions over 8 weeks (3 sessions per week), focusing on conventional physical therapy, cognitive training, and task-oriented exercises to enhance motor function and cognitive abilities. This group serves as a comparison to evaluate the effectiveness of VR-based rehabilitation. Neurophysiological changes will be monitored using EEG, MRI, and motion analysis to assess functional improvements.
  Arms: Active Control Group

SUMMARY:
This randomized controlled trial (RCT) evaluates the effectiveness of virtual reality (VR) rehabilitation in improving cognitive, emotional, social, and motor functions in patients with neurological disorders (ABI, SCI, MS, PD). It investigates whether VR improves motor and cognitive functions more than traditional therapy, identifies neurophysiological changes (EEG, fNIRS, MRI), and assesses the integration of VR with NIBS or telerehabilitation. Conducted over three years at IRCCS Centro Neurolesi Bonino Pulejo, participants are randomly assigned to either a VR training group or an active control group receiving traditional rehabilitation. Procedures include baseline assessments (T0), 20 rehabilitation sessions over 8 weeks, post-intervention evaluations (T1), and a 3-month follow-up (T2). Primary outcomes measure motor and cognitive function (MoCA, MMSE, FIM, TUG, Berg Balance Scale), neurophysiological changes (EEG, MRI, fNIRS, motion analysis), and emotional/social function (Empathy Quotient, Hamilton Depression Scale).

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) aims to evaluate the effectiveness of virtual reality (VR) rehabilitation in improving cognitive, emotional, social, and motor functions in patients with neurological and neurodegenerative disorders (Acquired Brain Injuries, Spinal Cord Injuries, Multiple Sclerosis, and Parkinson's Disease). The study also explores neurophysiological changes and the potential benefits of combining VR with non-invasive brain stimulation (NIBS) and telerehabilitation.

Objectives:

Primary Objectives:

Assess the effectiveness of VR-based rehabilitation in enhancing cognitive and motor functions.

Identify neurophysiological changes (EEG, fNIRS, MRI) associated with functional recovery.

Secondary Objectives:

Identify behavioral and neurophysiological biomarkers predictive of rehabilitation outcomes.

Compare the effectiveness of different VR devices for rehabilitation. Evaluate the impact of VR telerehabilitation on recovery and continuity of care.

Explore the synergistic effects of VR combined with NIBS.

Methods:

Study Site: IRCCS Centro Neurolesi Bonino Pulejo. Duration: 3 years. Participants: 328 individuals with neurological disorders (18-75 years old).

Design:

Participants will be randomized into two groups:

VR Training Group: Engages in immersive VR-based rehabilitation. Active Control Group: Receives conventional therapy. Sessions: 20 sessions over 8 weeks (3 times per week).

Assessments at 3 time points:

T0 (Baseline): Neurological, neuropsychological, motor, and neurophysiological evaluations.

T1 (Post-intervention): Repeat assessments to measure immediate effects. T2 (Follow-up at 3 months): Evaluate the maintenance of improvements.

Assessments & Outcome Measures:

Cognitive Function: MoCA, MMSE, ACE-R, Rao's Battery. Motor Function: Functional Independence Measure (FIM), TUG, Tinetti Scale, Berg Balance Scale.

Neurophysiological Changes: EEG, fNIRS, MRI, eye-tracking, motion analysis, sEMG.

Emotional & Social Function: Short Empathy Quotient (EQ-short), Faux Pas Test, Hamilton Depression Scale.

Usability & Acceptance: System Usability Scale (SUS).

Expected Impact:

This study aims to advance personalized rehabilitation strategies, improve accessibility to innovative therapies (e.g., telerehabilitation), and optimize the use of VR-based interventions in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years
* Diagnosis:

Parkinson's Disease (PD) (MDS Clinical Diagnostic Criteria) Multiple Sclerosis (MS) (McDonald Criteria) Spinal Cord Injury (SCI) (ASIA Impairment Scale) Acquired Brain Injury (ABI) (WHO Criteria for Stroke)

* Education: Minimum of 5 years of formal education
* Cognitive and physical ability to engage in rehabilitation

Exclusion Criteria:

* Major psychiatric disorders (e.g., psychosis, severe depression, anxiety disorders)
* Severe medical conditions that impair participation
* Sensory or motor impairments preventing VR interaction
* Contraindications for MRI (e.g., pacemakers, incompatible implants)
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2025-01-16 (Actual); Primary Completion 2027-09-29 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Cognitive Function | Baseline (T0), Post-Intervention (T1: 8 weeks), and Follow-Up (T2: 3 months post-intervention).
  Change in cognitive function from baseline (T0) to post-intervention (T1) and follow-up at 3 months (T2), assessed through standardized neuropsychological tests (Montreal Cognitive Assessment - MOCA). A clinically significant improvement is defined as a measurable increase in at least two subscales of the respective cognitive tests.
Improvement in Motor Function | Baseline (T0), Post-Intervention (T1: 8 weeks), and Follow-Up (T2: 3 months post-intervention).
  Change in motor function from baseline (T0) to post-intervention (T1) and follow-up at 3 months (T2), assessed through standardized clinical tests, including the Berg Balance Scale. A clinically significant improvement is defined as a measurable increase in functional mobility and balance scores.

SECONDARY OUTCOMES:
Neurophysiological Changes Associated with Rehabilitation | Baseline (T0), Post-Intervention (T1: 8 weeks), and Follow-Up (T2: 3 months post-intervention).
  Change in neurophysiological markers from baseline (T0) to post-intervention (T1) and follow-up (T2), assessed through EEG. Significant changes will be identified based on increased functional connectivity and structural adaptations indicative of neuroplasticity.
Effectiveness of Telerehabilitation | Baseline (T0), Post-Intervention (T1: 8 weeks), and Follow-Up (T2: 3 months post-intervention)
  Comparison of functional improvements between participants receiving VR-based rehabilitation in clinical settings versus those undergoing a telerehabilitation protocol. Changes in motor and cognitive function will be assessed from baseline (T0) to post-intervention (T1) and follow-up (T2) using MoCA. Accessibility, adherence, and patient-reported outcomes will also be analyzed to evaluate the feasibility and effectiveness of remote VR-based rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Maggio, PhD, PsyD, Principal Investigator — IRCCS Centro Neurolesi Bonino Pulejo
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Italy/Me, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD related to primary and secondary outcome measures will be shared. This includes data on cognitive performance, social cognition, neurophysiological parameters (EEG and MRI biomarkers), gait analysis, and eye movement metrics. Data will be made available to qualified researchers upon reasonable request, following ethical and legal guidelines to ensure participant confidentiality. Access will be provided through a secure platform for a limited period after the study's completion. Specific requests will be evaluated on a case-by-case basis, and approved researchers must agree to terms of use.
Supporting Information: SAP
Time Frame: IPD and supporting documentation, including the Statistical Analysis Plan (SAP), will be available starting 6 months after the study's primary completion date. Access will be provided for 5 years from the initial availability date, ensuring adequate time for secondary analyses while maintaining relevance to ongoing research efforts.
Access Criteria: Requests for access to Individual Participant Data (IPD) and supporting documentation will be evaluated by the study's data-sharing committee. Researchers must submit a proposal detailing their study objectives, statistical analysis plans, and ethical approval. Access will be granted for scientifically valid purposes, following a signed data use agreement. Requests should be directed to: mariagrazia.maggio@irccsme.it.

REFERENCES:
- [Background] Maggio MG, Maresca G, De Luca R, Stagnitti MC, Porcari B, Ferrera MC, Galletti F, Casella C, Manuli A, Calabro RS. The Growing Use of Virtual Reality in Cognitive Rehabilitation: Fact, Fake or Vision? A Scoping Review. J Natl Med Assoc. 2019 Aug;111(4):457-463. doi: 10.1016/j.jnma.2019.01.003. Epub 2019 Feb 8. PMID 30739728
- [Background] De Luca R, Russo M, Naro A, Tomasello P, Leonardi S, Santamaria F, Desiree L, Bramanti A, Silvestri G, Bramanti P, Calabro RS. Effects of virtual reality-based training with BTs-Nirvana on functional recovery in stroke patients: preliminary considerations. Int J Neurosci. 2018 Sep;128(9):791-796. doi: 10.1080/00207454.2017.1403915. Epub 2018 Feb 2. PMID 29148855
- [Background] Maggio MG, Bonanno M, Manuli A, Onesta MP, De Luca R, Quartarone A, Calabro RS. Do Individuals with Spinal Cord Injury Benefit from Semi-Immersive Virtual Reality Cognitive Training? Preliminary Results from an Exploratory Study on an Underestimated Problem. Brain Sci. 2023 Jun 13;13(6):945. doi: 10.3390/brainsci13060945. PMID 37371423